CLINICAL TRIAL: NCT07187908
Title: A Multicenter, Exploratory Clinical Study of Efbemalenograstim Alfa-vuxw Injection for Primary/Secondary Prevention in Patients With Solid Tumors at High Risk for Febrile Neutropenia (FN) or Intermediate Risk of Chemotherapy Regimens Associated With Other Risk Factors in FN
Brief Title: Efbemalenograstim Alfa for Primary/Secondary Prevention in Patients With Solid Tumors at High Risk for Febrile Neutropenia (FN) or Intermediate Risk of Chemotherapy Regimens Associated With Other Risk Factors in FN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: West China Hospital (Other)
Responsible Party: Principal Investigator, Zhenzhen Liu, Director, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Guard-001
Record Dates: First submitted 2025-04-22; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Primary/Secondary Prevention; High Risk for Febrile Neutropenia of Chemotherapy Regimens; Intermediate Risk of Chemotherapy Regimens Associated With Other Risk Factors in Febrile Neutropenia
Keywords: Efbemalenograstim alfa; primary/secondary prevention; febrile neutropenia of chemotherapy regimens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treated with Efbemalenograstim alfa for primary/secondary prevention after the chemotherapy (Experimental)
  Interventions: Drug: Efbemalenograstim alfa Injection

INTERVENTIONS:
Drug: Efbemalenograstim alfa Injection — The patients with solid tumor who were at high risk for febrile neutropenia or intermediate risk of chemotherapy regimens associated with other risk factors in febrile neutropenia would be injected Efbemalenograstim alfa for primary/secondary prevention.

SUMMARY:
Efbemalenograstim alfa for primary/secondary prevention in patients with solid tumors at high risk for febrile neutropenia (FN) or Intermediate risk of chemotherapy regimens associated with other risk factors in FN

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign the informed consent form and be able to comply with the requirements of the protocol;
* Age≥ 18 years old, ≤ 75 years old;
* Patients with solid tumors confirmed by histopathology or cytology;
* Cohort 1 requires that the patient has not used G-CSF drugs during this chemotherapy treatment;
* Cohort 2 requires patients to suffer ≥3 grade ANC reduction after the first course of chemotherapy, and there still has the risk in the subsequent chemotherapy;
* Patients planned to receive at least 2 courses of chemotherapy regimens with FN high risk or Intermediate risk with other risk factors (including, but not limited to,≥65 years-old, poor nutritional/performance status i.e., ECOG score ≥2, etc.);
* ECOG score 0-2;
* Expected survival of not less than 12 weeks;
* Neutrophil count (ANC) ≥ 2.0×109/L, hemoglobin (Hb) ≥90g/L and platelet (PLT) ≥80 × 109/L before enrollment;
* Liver and kidney function meet the following criteria: total bilirubin ≤ 1.5 times the upper limit of normal, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of normal, serum creatinine ≤ 1.5 times the upper limit of normal;
* Left Ventricular Ejection Fractions≥50%;
* Women of non-childbearing potential, i.e. women who have been postmenopausal for at least 1 year or have undergone sterilization surgery (bilateral tubal ligation, double oophorectomy or hysterectomy); Patients of childbearing potential agree to use adequate contraception within 1 month prior to the start of the trial and 30 days after the end of the study: condoms, spermicidal condoms, foams, gels, diaphragms, intrauterine devices (IUDs), contraceptives (administered orally or by injection).
* The investigator judges that the patient can tolerate treatment with Efbemalenograstim alfa.

Exclusion Criteria:

* Uncontrolled infection within 72 hours prior to chemotherapy or receiving systemic antibiotic therapy;
* Pregnant or lactating women;
* Have received bone marrow transplantation or stem cell transplantation in the past;
* Have 2 or more kinds of primary malignant tumors at the same time; However, the following exceptions are: 1) malignant tumors that have complete response for at least 2 years prior to enrollment and do not require other treatment during the study period; 2) non-melanoma skin cancer or lentigo maligna that has been adequately treated and has no evidence of disease recurrence; 3) carcinoma in situ that has been adequately treated and has no evidence of disease recurrence;
* Psychiatric or brain metastases;
* Surgical procedure and/or presence of trauma within 4 weeks;
* Clinical, electrocardiogram or other means of diagnosis of acute congestive heart failure, cardiomyopathy or myocardial infarction;
* Concomitant diseases that may lead to splenomegaly;
* Subjects with diagnosis of acute infection, chronic active hepatitis B within 1 year (unless known to be negative for hepatitis B virus antigen prior to enrollment), or hepatitis C;
* Known human immunodeficiency virus (HIV) seropositive, or AIDS;
* Active tuberculosis disease; or recent exposure to a person with tuberculosis, unless the tuberculin test is negative; or tuberculosis patients receiving treatment; or chest x-ray for suspected cases of tuberculosis;
* Patients with sickle cell anemia;
* Known hypersensitivity to granulocyte colony-stimulating factors or excipients of drugs;
* Use of other research drugs of the same type within 1 month before being selected for this study;
* In the opinion of the investigator, the patient has diseases or symptoms that are not suitable for participation in this study, and the study drug may harm the patient's health or affect the judgment of adverse events.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1076 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Incidence of ≥3 grade ANC reduction in patients after primary prevention with Efbemalenograstim alfa after the 1st cycle of chemotherapy | Evaluate the incidence of grade ≥3 ANC at the end of Cycle 1 (Cycle 1 is 21 days)
Cohort 2: Incidence of ≥3 grade ANC reduction in patients after secondary prevention with Efbemalenograstim alfa after the 2nd cycle of chemotherapy | Evaluate the incidence of grade ≥3 ANC at the end of Cycle 2 (Cycle 2 is 21 days)

SECONDARY OUTCOMES:
Incidence of febrile neutropenia (FN) of each cycle of chemotherapy | At the end of each cycle(each cycle is 21 days), an average of 3 months
Cohort 1: Incidence of ≥3 grade ANC reduction in patients after primary prevention with Efbemalenograstim alfa after the 2nd/3rd/4th cycle of chemotherapy | At the end of Cycle 2, 3 and 4 (each cycle is 21 days)
Cohort 2: Incidence of ≥3 grade ANC reduction in patients after secondary prevention with Efbemalenograstim alfa after the 3rd/4th cycle of chemotherapy | At the end of Cycle 3, 4 (each cycle is 21 days)
Safety indicators | Through study completion and 1 month post-treatment, an average of 4 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Injectable antibiotic use rate in each chemotherapy cycle | During the treatment of chemotherapy, an average of 3 months
The per capita number of doses of G-CSF products in each chemotherapy cycle | During the treatment of chemotherapy, an average of 3 months
Incidence of chemotherapy dose reduction (10% ≥reduction in the dose of any chemotherapy drugs) and chemotherapy delay (≥ 2 days later than planned) due to neutropenia in each chemotherapy cycle | During the treatment of chemotherapy, an average of 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Henan cancer hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results will be shared